CLINICAL TRIAL: NCT03440710
Title: The Therapeutic Effect of Balloon Eustachian Tuboplasty (BET) in Chronic Otitis Media (COM) With Eustachian Tube Dysfunction (ETD)
Brief Title: The Therapeutic Effect of BET in COM With ETD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The Effect of BET in COM
Record Dates: First submitted 2018-02-11; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Balloon Eustachian Tuboplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with BET (Experimental): with BET and Tympanoplast
  Interventions: Procedure: BET
- without BET (Other): with Tympanoplast only
  Interventions: Procedure: BET

INTERVENTIONS:
Procedure: BET — Balloon Eustachian Tuboplasty

SUMMARY:
Currently, surgical treatment of patients with chronic otitis media is one of the most important treatment methods. However, the current results show that some patients with eustachian tube dysfunction can't reconstruct the gas-containing structure of the middle ear after operation.

This is a randomized controlled trial that aims to evaluate the therapeutic effect of balloon eustachian tuboplasty (BET) for the treatment in chronic otitis media (COM) with eustachian tube dysfunction (ETD). This future study will aim to address the question: Does BET gain better recovery of auditory function and lower recurrence rate in chronic otitis media with eustachian tube dysfunction?

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need tympanoplasty, with clear diagnosis of chronic otitis media, middle ear cholesteatoma;
2. Patients with eustachian tube dysfunction using TMM;
3. Subjects or their legal representatives can understand the purpose of the study, show sufficient compliance with the research protocol, and sign the informed consent form.

Exclusion Criteria:

1. Secondary chronic otitis media (after head and neck cancer radiotherapy);
2. Ipsilateral ear recurrence after surgical treatment, requiring secondary surgery;
3. Two tympanoplasty surgery;
4. Typical allergic rhinitis, nasal endoscopy or imaging studies suggest chronic rhinosinusitis, nasal polyps and other short-term eustachian tube function of a greater impact on the disease;
5. poor general health, with severe liver and kidney dysfunction, coagulation disorders, cardiovascular disease, neurological diseases can not tolerate surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate in chronic otitis media with eustachian tube dysfunction | 6months after the surgery
  Recurrence rate in chronic otitis media with eustachian tube dysfunction: with BET vs without BET

SECONDARY OUTCOMES:
Hearing change in chronic otitis media with eustachian tube dysfunction | before the surgery, and 6months after the surgery
  Hearing outcome in chronic otitis media with eustachian tube dysfunction: with BET vs without BET
The change of Eustachian tube function using TUBOMANOMETRY (TMM) | before the surgery, and 6months after the surgery
  Eustachian tube function before and after surgery using TUBOMANOMETRY (TMM)

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607